CLINICAL TRIAL: NCT02185573
Title: Evaluation of Two Different Methods of Resin Composite Application Using Bulk-fill Technique In Class II Restorations
Brief Title: Evaluation of Two Different Methods of Resin Composite Application In Class II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-OperDent-01-2014
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Class II Dental Restorations
Keywords: Bulk fill; SonicFill; resin composite application; class II restoration
MeSH Terms: interventions — Filtek Bulk Fill; SonicFill

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Technique (No Intervention): Multi-layer filling technique
- Bulk fill technique (Active Comparator): Bulk fill technique
  Interventions: Procedure: Bulk fill
- SonicFill technique (Experimental): SonicFill technique
  Interventions: Procedure: SonicFill

INTERVENTIONS:
Procedure: Bulk fill — This is one of the composite restoration application techniques
  Arms: Bulk fill technique
Procedure: SonicFill — This is the recent intervention under evaluation
  Arms: SonicFill technique

SUMMARY:
Three clinical groups will be evaluated. Each group of patients will undergo one method of Resin Composite application (multi-layer technique 'control group' - bulk-fill Technique - Sonicfill technique). The restored teeth will be followed-up till one year. A comparison is going to be made between the three groups in relation to the modified United Sates Public Health Service (USPHS) criteria of good restorations.

DETAILED DESCRIPTION:
The modified USPHS criteria include the evaluation of seven characteristics of the restorations: color match, marginal integrity, surface texture, wear of both restoration and antagonist, recurrent dental caries, fracture or detachment, and gingivitis around the abutment.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperated patients.
2. Good general health.
3. Good oral hygiene.
4. Aged 15 to 60 years.
5. Class II restoration (upper or lower)
6. Full erupted teeth.
7. Caries value D3 -D4 according to Daignodent.

Exclusion Criteria:

1. If the caries value according to Daignodent is less than D3 -D4.
2. If the tooth is partially erupted.
3. Class II box-like cavity only without any extensions.
4. Patient outside the required age range (15-60 years).
5. Bad oral hygiene.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Color Match | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Color match
  1. The restoration appears to match the shade and translucency of adjacent tooth tissues.
  2. The restoration does not match the shade and translucency of adjacent tooth tissues, but the mismatch is within the range of tooth shade.
  3. The restoration does not match the shade and translucency of adjacent tooth tissues, and the mismatch is outside the normal range of tooth shade and translucency.
Change in Marginal Integrity | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Marginal integrity
  1. The explorer does not catch when drawn across the surface of the restoration toward the tooth, or, if the explorer does catch, there is no visible crevice along the periphery of the restoration.
  2. The explorer catches and there is visible evidence of crevice, into which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure.
  3. the explorer penetrates a crevice defect.
Change in Surface Texture | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Surface texture:
  1. Surface texture is similar to polished enamel as determined by means of a sharp explorer.
  2. Surface texture is gritty similar to a surface subject to a white stone or similar to a composite containing supramicron sizes particles.
  3. Surface pitting is sufficiently coarse to inhibit the continuous movement of an explorer across the surface.
Change in Restoration Wear | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Wear
  1. The restoration is continuation of existing anatomic form or is slightly flattened.
  2. A surface concavity is evident.
  3. There is a loss of restorative substance such that a surface concavity is evident. Replacement or restorative treatment is required.
Recurrent dental caries | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Recurrent dental caries:
  1. The restoration is a continuation of existing anatomic form adjacent to the restoration.
  2. There is visual evidence of dark deep discoloration adjacent to the restoration.
The Fracture/detachment Status | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Fracture/detachment:
  1. No bulk fracture/detachment is present.
  2. Bulk fracture/ detachment is evident.
Change in gingival status | Assessment will be done at (T0) within the first hour following composite sitting, (T1) after 3 months, (T2) after six months, (T3) after six months, (T4) at 12 months following application.
  Gingival status
  1. No clinical inflammation is present.
  2. Clinical inflammation is present.

CONTACTS AND LOCATIONS:
Overall Officials: Rahaf Alkurdi, DDS MSc, Principal Investigator — PhD student, Department of Operative Dentistry, University of Damascus Dental School, Damascus; Souad Abboud, DDS MSc PhD, Study Director — Associate Professor, Operative Dentistry Department, University of Damascus Dental School, Damascus
Locations (1):
- Department of Operative Dentistry, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Manhart J, Hickel R. [Bulk-fill-composites. Modern application technique of direct composites for posterior teeth]. Swiss Dent J. 2014;124(1):19-37. doi: 10.61872/sdj-2014-01-02. French, German. PMID 24665478
- [Background] van Dijken JW, Pallesen U. A randomized controlled three year evaluation of "bulk-filled" posterior resin restorations based on stress decreasing resin technology. Dent Mater. 2014 Sep;30(9):e245-51. doi: 10.1016/j.dental.2014.05.028. Epub 2014 Jun 21. PMID 24958689
- [Background] Ching K. Deep and fast: Kerr's SonicFill bulk fill composite. HDA Now. 2012 Spring:24-5. No abstract available. PMID 22984718
- [Background] Furness A, Tadros MY, Looney SW, Rueggeberg FA. Effect of bulk/incremental fill on internal gap formation of bulk-fill composites. J Dent. 2014 Apr;42(4):439-49. doi: 10.1016/j.jdent.2014.01.005. Epub 2014 Jan 27. PMID 24480086
- [Background] Campos EA, Ardu S, Lefever D, Jasse FF, Bortolotto T, Krejci I. Marginal adaptation of class II cavities restored with bulk-fill composites. J Dent. 2014 May;42(5):575-81. doi: 10.1016/j.jdent.2014.02.007. Epub 2014 Feb 18. PMID 24561041